CLINICAL TRIAL: NCT01013558
Title: NO PAIN: New Options for Preoperative Anesthesia in Intrauterine Needling
Brief Title: New Options for Preoperative Anesthesia in Intrauterine Needling
Acronym: NO PAIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Leuven University Medical Center (Unknown)
Responsible Party: F.P.H.A. Vandenbussche, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04.014
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-11

CONDITIONS: Stress; Pain
Keywords: fetal pain; intrauterine; needling
MeSH Terms: conditions — Pain | interventions — Remifentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- remifentanil (Active Comparator)
  Interventions: Drug: Remifentanil
- saline (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Remifentanil — 0.15 microgram/kg/min continuous infusion.
  Arms: remifentanil
Drug: saline — continuous infusion
  Arms: saline

SUMMARY:
The concept of fetal pain is becoming increasingly relevant due to growing possibilities for invasive intrauterine treatment. There is much debate as to whether the fetus is mature enough to be able to perceive pain at all. Recent studies have suggested that the fetus is at least capable of exhibiting a stress response to intrauterine needling. Intrauterine transfusions are most commonly performed by inserting a needle either in the umbilical cord root at the placental surface, or in the intrahepatic portion of the umbilical vein of the fetus. Recently, intrauterine needling in the intrahepatic vein has been shown to result in alterations in fetal stress hormones, which has been interpreted as a reaction to pain. These changes were not observed in intrauterine needling in the umbilical cord root, or after administration of analgesics to the fetus. The investigators tested the hypothesis that remifentanil provides fetal analgesia, assessed by a reduced fetal stress response. The investigators performed a randomised controlled trial comparing fetal stress response between patients undergoing intrauterine transfusions for alloimmune fetal anemia receiving remifentanil, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* clinically indicated intrauterine transfusion
* red cell alloimmunisation

Exclusion Criteria:

* severe adipositas
* suspicion of structural anomalies
* fetal hydrops
* contraindication for remifentanil

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
evidence of fetal stress response by changes in fetal stress hormones beta-endorphin, noradrenalin and cortisol | 15-60 minutes

SECONDARY OUTCOMES:
influence of analgesics (remifentanil) on the fetal stress response | 15-60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Frank P.H.A. Vandenbussche, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Andrewartha K, Grivell RM. Perioperative pharmacological interventions for fetal immobilisation during fetal surgery and invasive procedures. Cochrane Database Syst Rev. 2022 May 13;5(5):CD011068. doi: 10.1002/14651858.CD011068.pub2. PMID 35553414